CLINICAL TRIAL: NCT04089202
Title: Comparing Electronic Versus In-Person Access to Specialty Diabetes Expertise
Brief Title: Diabetes eConsult Non-Inferiority Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll additional participants and funding ended.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-38363
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Diabetes
Keywords: Diabetes specialty care; Flash glucose monitoring; Clinical pharmacists; eConsults; Freestyle Libre sensor
MeSH Terms: conditions — Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- In-person visit arm (Active Comparator): In this arm, patients meeting eligibility criteria and consented into the study are randomized to an in-person visit with an Endocrinologist. This is currently the standard of care for patients referred for diabetes specialty care.
  Care by the Endocrinologist is provided as would typically be done, taking into account patient factors and preferences.
  Surveys will be administered to measure patient burden and self efficacy.
  Interventions: Other: Standard of care
- Freestyle Libre sensor arm (Experimental): In this arm, patients meeting eligibility criteria and consented into the study are randomized to have the Freestyle Libre Pro continuous glucose monitor (CGM) placed at their primary care clinic. The data collected from the diagnostic CGM will be utilized in conjunction with diet, exercise and medication logs provided by the patient and information from the patient's electronic medical record to complete an eConsult with treatment recommendations. Implementation of these recommendations will be per the primary care provider's discretion in conjunction with conversation with the patient in follow up visits.
  Surveys will be administered to measure patient burden and self efficacy.
  Interventions: Other: eConsult

INTERVENTIONS:
Other: eConsult — Completion of electronic consult utilizing data collected from flash glucose monitoring
  Arms: Freestyle Libre sensor arm
Other: Standard of care — Care by the Endocrinologist is provided as would typically be done, taking into account patient factors and preferences.
  Arms: In-person visit arm

SUMMARY:
Flash glucose monitoring is an FDA-approved and widely clinically available, glucose monitoring technology that is worn on the body and measures glucose values every 15 minutes, storing this data for up to 14 days. The Freestyle Libre Pro is already used as a diagnostic technology in clinical care. It provides a full 24-hour glucose profile for each day that the sensor is worn and that can be correlated with daily activities, medication administration, food intake, and other factors that are contextually relevant in meeting glycemic goals for an individual patient.

In this study, patients referred to Endocrinology for specialty diabetes care will be randomized to an in-person visit as is typically done or to wear the Freestyle Libre Pro placed by staff at their primary care clinic. Patients who wear the Freestyle Libre Pro will have a professional interpretation of their glucose data completed by an endocrinologist as well as a remote eConsult completed using this glucose data and information from their medical record. The recommendations from the eConsult regarding medication and lifestyle adjustment as well as potential referral on to see Endocrinology will be implemented by the primary care physician at their clinical discretion.

The investigators will utilize glycemic measures including hemoglobin A1c, number of clinical visits (outpatient, inpatient and emergency department) for diabetes care, patient reported outcomes including self-efficacy, and patient and provider assessments of burden to determine if eConsults utilizing flash glucose monitoring technology are non-inferior to in-person visits with a diabetes specialist.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 18-80, inclusive
* Diagnosed with type 2 diabetes at least 6 months prior to screening
* Not previously seen within the prior three years in the endocrinology clinic for diabetes management
* Referred to endocrinology for diabetes care directly from primary care
* Willing to wear an Abbott® FreeStyle Libre Pro for 7-14 days
* English speaking
* Able and willing to complete questionnaires

Exclusion Criteria:

* Planned travel or surgery during the time of libre wear
* Patients without a diagnosis of type 2 diabetes, including individuals with type 1 diabetes and gestational diabetes
* Women referred for diabetes care during pregnancy, or while breastfeeding or who intend to become pregnant during involvement in this trial
* Currently using real time CGM or FGM system
* Concurrent involvement in another clinical trial using diabetes pharmacotherapy
* Individuals with active malignancy undergoing treatment with chemotherapy and/or high dose glucocorticoids
* Individuals with rheumatic disease undergoing treatment with high dose glucocorticoids
* Planned magnetic resonance imaging (MRI), computed tomography (CT) scan, or high-frequency electrical heat (diathermy) treatment during the time of Libre wear
* Any cognitive or other disorders, in the investigator's opinion, that may interfere with participation or ability to follow the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c (A1c) at baseline | baseline
  A1c will be obtained as standard of care and values documented in the medical record.
Hemoglobin A1c (A1c) at 3 months | 3 months
  A1c will be obtained as standard of care and values documented in the medical record.
Hemoglobin A1c (A1c) at 6 months | 6 months
  A1c will be obtained as standard of care and values documented in the medical record.
Hemoglobin A1c (A1c) at 12 months | 12 months
  A1c will be obtained as standard of care and values documented in the medical record.
Percentage change in A1c to 6 months | baseline, 6 months
  The percent change in A1c will be calculated from baseline to six months
Percentage change in A1c to 12 months | baseline, 12 months
  The percent change in A1c will be calculated from baseline to 12 months
Proportion of patients with A1c <7% | 6 months, 12 months
  The proportion of participants with A1c <7% (ADA target) will be calculated.
Proportion of patients with A1c <8% | 6 months, 12 months
  The proportion of participants with A1c <8% (ADA target) will be calculated.
Glycemic control based on A1c | 12 months
  A1c reduction of > 1% with 20% non-inferiority margin

SECONDARY OUTCOMES:
Number of clinical visits for diabetes care | 12 months
  The number of clinical visits (outpatient, inpatient and emergency department) for diabetes care will be calculated for each participant
Patient assessment of care burden | within 2 weeks of the physician visit or eConsult
  Modified assessment of perceived research burden
Provider assessment of acceptability | at baseline, 6 months, and completion of study period
  Results from a 16 item post intervention questionnaire developed by the investigators will be used to assess provider acceptability. It includes 10 questions with a 5 item Likert scale from 1= Strongly disagree to 5= Strongly agree that asks about the usefulness, feasibility and how much they liked the eConsult and the physician visits. There are also 2 open-ended questions soliciting qualitative information about the intervention.
Patient self efficacy and disease burden based on diabetes self management questionnaire and problem areas in diabetes short five-item short form questionnaire | at baseline and 6 months
  Patient disease burden will be measured by the validated Problem Areas in Diabetes-5 question (PAID-5) survey. The five questions are from the original 20 item PAID survey (specifically questions 3, 6, 12, 16, and 19) and each has a 5-point Likert scale ranging from "not a problem" (score of 0) to "serious problem" (score of 4). The possible total scores of the PAID-5 ranges from 0 to 20, with higher scores implying greater emotional distress.
Efficacy of embedded clinical pharmacists | baseline, 3, 6, and 12 months
  Changes in hemoglobin A1c will be used to assess the efficacy of the embedded clinical pharmacists
Cost effectiveness analysis (CEA) | 12 months
  A Cost-Effectiveness Analysis will be done to compare the costs and health gains for the eConsult and standard of care interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Devin Steenkamp, MD, Principal Investigator — Boston Medical Center, Endocrinology, Diabetes & Nutrition
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No